CLINICAL TRIAL: NCT05306054
Title: Investigating the Associations Between Physical Activity, Knee Joint Loading and Joint Health Following Anterior Cruciate Ligament Reconstruction
Brief Title: Physical Activity, Knee Joint Loading and Joint Health
Status: Recruiting | Type: Observational
Sponsor: University of Bath (Other)
Collaborators: Versus Arthritis (Other)
Responsible Party: Principal Investigator, Karl Morgan, Chief Investigator, University of Bath
Other Study IDs: 304181
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Anterior Cruciate Ligament Injuries; Anterior Cruciate Ligament Rupture; Anterior Cruciate Ligament Tear; Post-traumatic Osteoarthritis; Anterior Cruciate Ligament Reconstruction
Keywords: Physical Activity; Knee Joint Loading; Cumulative Load; Biomarkers; Musculoskeletal Modelling; Patient Reported Outcomes
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood Serum and Plasma. Urine.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intra-Articular Knee Injury: Forty men and women aged 18-45 years old who are 1-7 years following an intra-articular knee injury.
- Controls: Forty men and women aged 18-45 years old who are matched to the injured group by age, sex and body mass index.

SUMMARY:
The purpose of this study is to investigate the association between time spent in moderate to vigorous physical activity and markers of cartilage metabolism in the years following anterior cruciate ligament reconstruction.

DETAILED DESCRIPTION:
Participants attend the laboratory on two or three occasions and wear accelerometers for the 10 days in between the first and second laboratory session. The first laboratory session involves urine sample collection, the completion of questionnaires, blood sample collection, acquisition of cross-sectional images of the thigh and calf, and a whole-body composition scan. The researchers will use the accelerometers at the wrist to measure time spent in moderate to vigorous physical activity, and the accelerometers at the ankle as an analogue for knee joint loading. The second laboratory session will consist of a 30-minute run on an instrumented treadmill (measures force of each step taken) whilst wearing non-invasive reflective markers, electromyography devices, and an accelerometer at the ankle. Participants are also invited to undergo optional repeated blood sampling to measure levels of markers of cartilage production and breakdown during rest and in response to a 30-minute run. If participants volunteer for the optional repeated blood sampling, they will be asked to attend a third laboratory session where blood samples will be taken at 24 hours after the run in the second laboratory session.

ELIGIBILITY:
Inclusion Criteria:

1. 18-39 years old (i.e., ≥18 and <40 years old)
2. Had an anterior cruciate ligament injury and reconstruction 1-7 years ago (i.e., ≥1 and ≤7 years ago)
3. Can have sustained damage to meniscus or cartilage, or sustained bone bruising when injured anterior cruciate ligament
4. Can participate regardless of the type of reconstruction surgery and if undergone meniscectomy
5. Completed anterior cruciate ligament reconstruction rehabilitation and either a surgeon, doctor or physiotherapist has provided clearance to participate in physical activity
6. Be able to attend the University of Bath within 2 hours of waking

Exclusion Criteria:

1. Had another significant knee injury either before, at the same time, or after the anterior cruciate ligament injury (e.g., if they injured another ligament in their knee or had a fracture or dislocation)
2. Injured the anterior cruciate ligament in both knees (bilateral ACL injury)
3. Have/are experiencing a musculoskeletal, cardiovascular, respiratory, immune, metabolic or neurological disease or disorder
4. Under 18 or over 39 (i.e., ≥40) years of age
5. Body Mass Index ≥40 kg/m²
6. Pregnancy
7. Positive responses to the Physical Activity Readiness Questionnaire (aside from any involved knee joint issues)

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young men and women who are aged 18-39 years old and are 1-7 years following their anterior cruciate ligament injury and surgery.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Ratio of urine concentration of c-telopeptide of type II collagen to serum concentration of c-propeptide of type II procollagen | Day 1
  Urine concentration of c-telopeptide of type II collagen (uCTX-II) is a marker of cartilage degradation. Serum concentration of c-propeptide of type II procollagen (sCP-II) is a marker of cartilage synthesis. The ratio between these two biomarkers as an indicator of knee joint health has previously been validated.

SECONDARY OUTCOMES:
Urine concentration of c-telopeptide of type II collagen | Day 1
  Urine concentration of c-telopeptide of type II collagen (uCTX-II) is a marker of cartilage degradation.
Serum concentration of c-propeptide of type II procollagen | Day 1
  Serum concentration of c-propeptide of type II procollagen (sCP-II) is a marker of cartilage synthesis.
Time spent in moderate to vigorous physical activity | Day 3-10
  Time spent in moderate to vigorous physical activity will be measured using GENEActiv accelerometers worn on the wrist. The devices have previously been validated to quantify physical activity domains.
Step count | Day 3-10
  Step count will be measured using GENEActiv accelerometers.
Knee joint reaction force | Day 11
  Knee joint reaction force will be measured using musculoskeletal modelling in OpenSim. We will use 3D motion capture to measure joint kinematics, an instrumented treadmill to measure ground reaction forces, and electromyography devices to measure muscle activation.
Cumulative knee joint reaction force | Days 3-11
  We are synchronising data collected by the GENEActiv tri-axial accelerometer with knee joint reaction force during walking and running. We then apply the relationship between these two variables (ascertained during the lab session) to the data collected during the 10 days of wear in free living to provide an estimation of cumulative knee joint reaction force.
Muscle cross-sectional area | Day 1
  We are using peripheral quantitative computerised tomography (pQCT) to measure muscle cross-sectional area. pQCT has previously been validated to measure muscle cross-sectional area.
Muscle density | Day 1
  We are using peripheral quantitative computerised tomography (pQCT) to measure muscle density. pQCT has previously been validated to measure muscle density.
Subcutaneous adipose tissue area | Day 1
  We are using peripheral quantitative computerised tomography (pQCT) to measure subcutaneous adipose tissue area. pQCT has previously been validated to measure subcutaneous adipose tissue area.
Intra-muscular fat content | Day 1
  We are using peripheral quantitative computerised tomography (pQCT) to measure intra-muscular fat content. pQCT has previously been validated to measure intra-muscular fat content.
Fat mass index | Day 1
  We are using dual-energy x-ray absorptiometry (DEXA) to measure fat mass index. DEXA has previously been validated to measure fat mass index.
Lean mass index | Day 1
  We are using dual-energy x-ray absorptiometry (DEXA) to measure lean mass index. DEXA has previously been validated to measure lean mass index.
Knee Injury and Osteoarthritis Outcome Score | Day 1
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) will be used to measure subjective knee joint health. It asks participants to report their symptoms (e.g., pain, stiffness) and function. The KOOS has been validated in a number of populations including those after knee injury.
Tampa Scale of Kinesiophobia - 11 score | Day 1
  The Tampa Scale of Kinesiophobia - 11 (TSK-11) will be used to measure fear of reinjury/movement. It has been validated in patients with musculoskeletal pain and in knee injury populations.
English Knee Self-Efficacy Scale score | Day 1
  The English Knee Self-Efficacy Scale (KSES-E) measures knee specific confidence during everyday tasks and physical activity. The KSES-E has been validated in knee injury populations.
Modified Godin Leisure Time Exercise Questionnaire score | Day 1
  The Modified Godin Leisure Time Exercise Questionnaire (GLTEQ) measures subjective physical activity over a typical seven day period.
Time spent in lower body resistance training per week | Day 1
  Time spent in lower body resistance training per week will be used to measure subjective time spent in lower body resistance training such as weights or body weight exercise.
Serum concentration of chondroitin sulphate 846 epitope | Day 11 and 12
  Serum concentration of chondroitin sulphate 846 epitope (sCS846) will be measured as marker of aggrecan synthesis.
Serum concentration of hyaluronic acid | Day 11 and 12
  Serum concentration of hyaluronic acid (HA) will be measured as marker of proteoglycan breakdown.

CONTACTS AND LOCATIONS:
Overall Officials: Karl Morgan, MSc, Principal Investigator — University of Bath
Locations (1):
- University of Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: No